CLINICAL TRIAL: NCT00562094
Title: Pantoprazole for the Treatment of GERD Associated Symptoms Focusing on Sleep Disorders.
Brief Title: Efficacy of Pantoprazole in Patients Older Than 12 Years With Reflux Associated Sleep Disorders (PULS)
Acronym: PULS
Status: Completed | Type: Observational
Sponsor: Nycomed (Industry)
Responsible Party: Medical Responsible, Nycomed Deutschland GmbH
Other Study IDs: PAN 20/40 PULS 07/10
Record Dates: First submitted 2007-11-12; First posted 2007-11-21 (Estimated); Results first posted 2010-09-24 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Erosive Gastroesophageal Reflux Disease; Non-Erosive Reflux Disease
Keywords: Pantoprazole; eGERD (Erosive Gastroesophageal Reflux Disease); NERD (Non-Erosive Reflux Disease); sleep disorders
MeSH Terms: conditions — Non-Erosive Reflux Disease; Sleep Wake Disorders | interventions — Pantoprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pantoprazole
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — This was an observational study. Therefore, the physician decided about dosage according to individual needs.

SUMMARY:
The aim of the study was to evaluate the effect of Pantoprazole 20 mg/40 mg for 14 days on symptoms in patients with NERD (non-erosive reflux disease) or eGERD (erosive gastroesophageal reflux disease) with special focus on the reduction of symptomatic sleep disorders.

ELIGIBILITY:
Main inclusion criteria:

* GERD
* NERD

Main exclusion criteria:

* Criteria as defined in the Summary of Product Characteristics

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients
Sampling Method: Non-Probability Sample
Enrollment: 8616 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Thomas D. Bethke, MD, MBA, Study Director — Nycomed Deutschland GmbH, 78467 Konstanz, Germany
Locations (840):
- Germany (840):
  - Nycomed Deutschland GmbH, Aachen
  - Nycomed Deutschland GmbH, Aalen
  - Nycomed Deutschland GmbH, Achern
  - Nycomed Deutschland GmbH, Achim
  - Nycomed Deutschland GmbH, Adenau
  - Nycomed Deutschland GmbH, Adorf
  - Nycomed Deutschland GmbH, Ahrensburg
  - Nycomed Deutschland GmbH, Aicha
  - Nycomed Deutschland GmbH, Albstadt
  - Nycomed Deutschland GmbH, Alfhausen
  - Nycomed Deutschland GmbH, Alpen
  - Nycomed Deutschland GmbH, Alpenrod
  - Nycomed Deutschland GmbH, Altenburg
  - Nycomed Deutschland GmbH, Altenholz
  - Nycomed Deutschland GmbH, Altenkirchen
  - Nycomed Deutschland GmbH, Alzenau in Unterfranken
  - Nycomed Deutschland GmbH, Alzey
  - Nycomed Deutschland GmbH, Amberg
  - Nycomed Deutschland GmbH, Angermünde
  - Nycomed Deutschland GmbH, Anklam
  - Nycomed Deutschland GmbH, Annaberg-Buchholz
  - Nycomed Deutschland GmbH, Annweiler am Trifels
  - Nycomed Deutschland GmbH, Apolda
  - Nycomed Deutschland GmbH, Arnsberg
  - Nycomed Deutschland GmbH, Arnsdorf
  - Nycomed Deutschland GmbH, Ascheberg
  - Nycomed Deutschland GmbH, Aschendorf
  - Nycomed Deutschland GmbH, Aschersleben
  - Nycomed Deutschland GmbH, Attenkirchen
  - Nycomed Deutschland GmbH, Aue
  - Nycomed Deutschland GmbH, Auerbach
  - Nycomed Deutschland GmbH, Augsburg
  - Nycomed Deutschland GmbH, Augustusburg
  - Nycomed Deutschland GmbH, Aumühle
  - Nycomed Deutschland GmbH, Babenhausen
  - Nycomed Deutschland GmbH, Bad Aibling
  - Nycomed Deutschland GmbH, Bad Bederkesa
  - Nycomed Deutschland GmbH, Bad Berka
  - Nycomed Deutschland GmbH, Bad Bevensen
  - Nycomed Deutschland GmbH, Bad Bramstedt
  - Nycomed Deutschland GmbH, Bad Buchau
  - Nycomed Deutschland GmbH, Bad Doberan
  - Nycomed Deutschland GmbH, Bad Dürkheim
  - Nycomed Deutschland GmbH, Bad Dürrheim
  - Nycomed Deutschland GmbH, Bad Essen
  - Nycomed Deutschland GmbH, Bad Fallingbostel
  - Nycomed Deutschland GmbH, Bad Klosterlausnitz
  - Nycomed Deutschland GmbH, Bad Kreuznach
  - Nycomed Deutschland GmbH, Bad Krozingen
  - Nycomed Deutschland GmbH, Bad Langensalza
  - Nycomed Deutschland GmbH, Bad Lauterberg im Harz
  - Nycomed Deutschland GmbH, Bad Liebenwerda
  - Nycomed Deutschland GmbH, Bad Lippspringe
  - Nycomed Deutschland GmbH, Bad Nauheim
  - Nycomed Deutschland GmbH, Bad Neustadt an der Saale
  - Nycomed Deutschland GmbH, Bad Oeynhausen
  - Nycomed Deutschland GmbH, Bad Oldesloe
  - Nycomed Deutschland GmbH, Bad Salzuflen
  - Nycomed Deutschland GmbH, Bad Sassendorf
  - Nycomed Deutschland GmbH, Bad Schussenried
  - Nycomed Deutschland GmbH, Bad Suderode
  - Nycomed Deutschland GmbH, Bad Tölz
  - Nycomed Deutschland GmbH, Bad Vilbel
  - Nycomed Deutschland GmbH, Bad Waldsee
  - Nycomed Deutschland GmbH, Bad Windsheim
  - Nycomed Deutschland GmbH, Baden-Baden
  - Nycomed Deutschland GmbH, Bahrdorf
  - Nycomed Deutschland GmbH, Bakum
  - Nycomed Deutschland GmbH, Balingen
  - Nycomed Deutschland GmbH, Ballenstedt
  - Nycomed Deutschland GmbH, Bamberg
  - Nycomed Deutschland GmbH, Bammental
  - Nycomed Deutschland GmbH, Barmstedt
  - Nycomed Deutschland GmbH, Bausendorf
  - Nycomed Deutschland GmbH, Bautzen
  - Nycomed Deutschland GmbH, Bechhofen
  - Nycomed Deutschland GmbH, Beeskow
  - Nycomed Deutschland GmbH, Bergisch Gladbach
  - Nycomed Deutschland GmbH, Bergkamen
  - Nycomed Deutschland GmbH, Bergtheim
  - Nycomed Deutschland GmbH, Berlin
  - Nycomed Deutschland GmbH, Bernburg
  - Nycomed Deutschland GmbH, Berne
  - Nycomed Deutschland GmbH, Bernkastel-Kues
  - Nycomed Deutschland GmbH, Beucha
  - Nycomed Deutschland GmbH, Beverungen
  - Nycomed Deutschland GmbH, Biberach
  - Nycomed Deutschland GmbH, Bielefeld
  - Nycomed Deutschland GmbH, Bietigheim-Bissingen
  - Nycomed Deutschland GmbH, Birkenfeld
  - Nycomed Deutschland GmbH, Birkenwerder
  - Nycomed Deutschland GmbH, Bischofswerda
  - Nycomed Deutschland GmbH, Bitburg
  - Nycomed Deutschland GmbH, Blankenhain
  - Nycomed Deutschland GmbH, Blaustein
  - Nycomed Deutschland GmbH, Bochum
  - Nycomed Deutschland GmbH, Bodman-Ludwigshafen
  - Nycomed Deutschland GmbH, Bohmte
  - Nycomed Deutschland GmbH, Bonn
  - Nycomed Deutschland GmbH, Bonndorf
  - Nycomed Deutschland GmbH, Borna
  - Nycomed Deutschland GmbH, Bottendorf
  - Nycomed Deutschland GmbH, Bottrop
  - Nycomed Deutschland GmbH, Bovenden
  - Nycomed Deutschland GmbH, Börnsen
  - Nycomed Deutschland GmbH, Brake
  - Nycomed Deutschland GmbH, Brakel
  - Nycomed Deutschland GmbH, Bramsche
  - Nycomed Deutschland GmbH, Brand-Erbisdorf
  - Nycomed Deutschland GmbH, Braunsbedra
  - Nycomed Deutschland GmbH, Braunschweig
  - Nycomed Deutschland GmbH, Bredstedt
  - Nycomed Deutschland GmbH, Breidenbach
  - Nycomed Deutschland GmbH, Breitenfelde
  - Nycomed Deutschland GmbH, Bremen
  - Nycomed Deutschland GmbH, Bremerhaven
  - Nycomed Deutschland GmbH, Bretten
  - Nycomed Deutschland GmbH, Brilon
  - Nycomed Deutschland GmbH, Bröckel
  - Nycomed Deutschland GmbH, Brüel
  - Nycomed Deutschland GmbH, Brühl
  - Nycomed Deutschland GmbH, Buchloe
  - Nycomed Deutschland GmbH, Buckow
  - Nycomed Deutschland GmbH, Burg
  - Nycomed Deutschland GmbH, Burgbrohl
  - Nycomed Deutschland GmbH, Burgdorf, Hanover
  - Nycomed Deutschland GmbH, Burgsinn
  - Nycomed Deutschland GmbH, Burgstädt
  - Nycomed Deutschland GmbH, Burkardroth
  - Nycomed Deutschland GmbH, Burladingen
  - Nycomed Deutschland GmbH, Butzbach
  - Nycomed Deutschland GmbH, Büchen
  - Nycomed Deutschland GmbH, Büchenbach
  - Nycomed Deutschland GmbH, Bühlertann
  - Nycomed Deutschland GmbH, Castrop-Rauxel
  - Nycomed Deutschland GmbH, Celle
  - Nycomed Deutschland GmbH, Chemnitz
  - Nycomed Deutschland GmbH, Clausthal-Zellerfeld
  - Nycomed Deutschland GmbH, Claußnitz
  - Nycomed Deutschland GmbH, Cochem
  - Nycomed Deutschland GmbH, Coesfeld
  - Nycomed Deutschland GmbH, Cologne
  - Nycomed Deutschland GmbH, Coswig
  - Nycomed Deutschland GmbH, Cottbus
  - Nycomed Deutschland GmbH, Crimmitschau
  - Nycomed Deutschland GmbH, Crostwitz
  - Nycomed Deutschland GmbH, Cuxhaven
  - Nycomed Deutschland GmbH, Dachau
  - Nycomed Deutschland GmbH, Dargun
  - Nycomed Deutschland GmbH, Darmstadt
  - Nycomed Deutschland GmbH, Deggingen
  - Nycomed Deutschland GmbH, Deidesheim
  - Nycomed Deutschland GmbH, Delitzsch
  - Nycomed Deutschland GmbH, Denkendorf
  - Nycomed Deutschland GmbH, Denzlingen
  - Nycomed Deutschland GmbH, Dessau
  - Nycomed Deutschland GmbH, Detmold
  - Nycomed Deutschland GmbH, Dettmannsdorf
  - Nycomed Deutschland GmbH, Diepholz
  - Nycomed Deutschland GmbH, Dierdorf
  - Nycomed Deutschland GmbH, Dillingen
  - Nycomed Deutschland GmbH, Dillingen-Diefflen
  - Nycomed Deutschland GmbH, Dingolfing
  - Nycomed Deutschland GmbH, Dinkelsbühl
  - Nycomed Deutschland GmbH, Dinkelscherben
  - Nycomed Deutschland GmbH, Dinslaken
  - Nycomed Deutschland GmbH, Doberschütz
  - Nycomed Deutschland GmbH, Donaueschingen
  - Nycomed Deutschland GmbH, Dorsten
  - Nycomed Deutschland GmbH, Dortmund
  - Nycomed Deutschland GmbH, Döbeln
  - Nycomed Deutschland GmbH, Dörentrup
  - Nycomed Deutschland GmbH, Dörpen
  - Nycomed Deutschland GmbH, Dörzbach
  - Nycomed Deutschland GmbH, Dresden
  - Nycomed Deutschland GmbH, Dresden-Cossebaude
  - Nycomed Deutschland GmbH, Dudenhofen
  - Nycomed Deutschland GmbH, Duderstadt
  - Nycomed Deutschland GmbH, Duisburg
  - Nycomed Deutschland GmbH, Durach
  - Nycomed Deutschland GmbH, Düren
  - Nycomed Deutschland GmbH, Dürrröhrsdorf
  - Nycomed Deutschland GmbH, Düsseldorf
  - Nycomed Deutschland GmbH, Ebeleben
  - Nycomed Deutschland GmbH, Eberbach
  - Nycomed Deutschland GmbH, Eckernförde
  - Nycomed Deutschland GmbH, Edenkoben
  - Nycomed Deutschland GmbH, Ehingen
  - Nycomed Deutschland GmbH, Ehra-Lessien
  - Nycomed Deutschland GmbH, Ehrenkirchen
  - Nycomed Deutschland GmbH, Eilenburg
  - Nycomed Deutschland GmbH, Eimsheim
  - Nycomed Deutschland GmbH, Einbeck
  - Nycomed Deutschland GmbH, Eisenhüttenstadt
  - Nycomed Deutschland GmbH, Eiterfeld
  - Nycomed Deutschland GmbH, Ellhofen
  - Nycomed Deutschland GmbH, Ellwangen
  - Nycomed Deutschland GmbH, Elmshorn
  - Nycomed Deutschland GmbH, Elsenfeld
  - Nycomed Deutschland GmbH, Emmendingen
  - Nycomed Deutschland GmbH, Emsdetten
  - Nycomed Deutschland GmbH, Engelskirchen
  - Nycomed Deutschland GmbH, Ennepetal
  - Nycomed Deutschland GmbH, Eppelheim
  - Nycomed Deutschland GmbH, Erfurt
  - Nycomed Deutschland GmbH, Erkner
  - Nycomed Deutschland GmbH, Erlangen
  - Nycomed Deutschland GmbH, Eschelbronn
  - Nycomed Deutschland GmbH, Eschwege
  - Nycomed Deutschland GmbH, Eschweiler
  - Nycomed Deutschland GmbH, Essen
  - Nycomed Deutschland GmbH, Esslingen am Neckar
  - Nycomed Deutschland GmbH, Ettlingen
  - Nycomed Deutschland GmbH, Extertal
  - Nycomed Deutschland GmbH, Falkensee
  - Nycomed Deutschland GmbH, Feldafing
  - Nycomed Deutschland GmbH, Felsberg
  - Nycomed Deutschland GmbH, Feuchtwangen
  - Nycomed Deutschland GmbH, Finsterwalde
  - Nycomed Deutschland GmbH, Flensburg
  - Nycomed Deutschland GmbH, Floh-Seligenthal
  - Nycomed Deutschland GmbH, Flonheim
  - Nycomed Deutschland GmbH, Flöha
  - Nycomed Deutschland GmbH, Flörsheim-Dalsheim
  - Nycomed Deutschland GmbH, Forbach
  - Nycomed Deutschland GmbH, Föhren
  - Nycomed Deutschland GmbH, Frankenberg
  - Nycomed Deutschland GmbH, Frankenthal
  - Nycomed Deutschland GmbH, Frankfurt
  - Nycomed Deutschland GmbH, Freiburg im Breisgau
  - Nycomed Deutschland GmbH, Freinsheim
  - Nycomed Deutschland GmbH, Freising
  - Nycomed Deutschland GmbH, Freital
  - Nycomed Deutschland GmbH, Freudenstadt
  - Nycomed Deutschland GmbH, Freyung
  - Nycomed Deutschland GmbH, Friedland
  - Nycomed Deutschland GmbH, Friedrichsdorf
  - Nycomed Deutschland GmbH, Friedrichshafen
  - Nycomed Deutschland GmbH, Friedrichsthal
  - Nycomed Deutschland GmbH, Friesenheim
  - Nycomed Deutschland GmbH, Friolzheim
  - Nycomed Deutschland GmbH, Frohburg
  - Nycomed Deutschland GmbH, Furth im Wald
  - Nycomed Deutschland GmbH, Fürstenberg
  - Nycomed Deutschland GmbH, Fürstenwalde
  - Nycomed Deutschland GmbH, Fürth
  - Nycomed Deutschland GmbH, Gaggenau
  - Nycomed Deutschland GmbH, Garbsen
  - Nycomed Deutschland GmbH, Garmisch-Partenkirchen
  - Nycomed Deutschland GmbH, Geilenkirchen
  - Nycomed Deutschland GmbH, Gelnhausen
  - Nycomed Deutschland GmbH, Gelsenkirchen
  - Nycomed Deutschland GmbH, Gemünden
  - Nycomed Deutschland GmbH, Genthin
  - Nycomed Deutschland GmbH, Gera
  - Nycomed Deutschland GmbH, Gerbstedt
  - Nycomed Deutschland GmbH, Geretsried
  - Nycomed Deutschland GmbH, Geringswalde
  - Nycomed Deutschland GmbH, Germering
  - Nycomed Deutschland GmbH, Gernrode
  - Nycomed Deutschland GmbH, Gerstungen
  - Nycomed Deutschland GmbH, Gifhorn
  - Nycomed Deutschland GmbH, Gladbeck
  - Nycomed Deutschland GmbH, Gleichen
  - Nycomed Deutschland GmbH, Glinde
  - Nycomed Deutschland GmbH, Glindow
  - Nycomed Deutschland GmbH, Gnoien
  - Nycomed Deutschland GmbH, Gomaringen
  - Nycomed Deutschland GmbH, Gommern
  - Nycomed Deutschland GmbH, Gornau
  - Nycomed Deutschland GmbH, Gorxheimertal
  - Nycomed Deutschland GmbH, Goslar
  - Nycomed Deutschland GmbH, Görlitz
  - Nycomed Deutschland GmbH, Göttingen
  - Nycomed Deutschland GmbH, Gößnitz
  - Nycomed Deutschland GmbH, Gransee
  - Nycomed Deutschland GmbH, Grasleben
  - Nycomed Deutschland GmbH, Gräfinau-Angstedt
  - Nycomed Deutschland GmbH, Greifswald
  - Nycomed Deutschland GmbH, Greiz
  - Nycomed Deutschland GmbH, Grevesmühlen
  - Nycomed Deutschland GmbH, Grimma
  - Nycomed Deutschland GmbH, Grimmen
  - Nycomed Deutschland GmbH, Groitzsch
  - Nycomed Deutschland GmbH, Großaitingen
  - Nycomed Deutschland GmbH, Großbottwar
  - Nycomed Deutschland GmbH, Großefehn
  - Nycomed Deutschland GmbH, Großenehrich
  - Nycomed Deutschland GmbH, Großräschen
  - Nycomed Deutschland GmbH, Großschönau
  - Nycomed Deutschland GmbH, Gröden
  - Nycomed Deutschland GmbH, Grömitz
  - Nycomed Deutschland GmbH, Grundau
  - Nycomed Deutschland GmbH, Gundelsheim
  - Nycomed Deutschland GmbH, Gunzenhausen
  - Nycomed Deutschland GmbH, Güglingen
  - Nycomed Deutschland GmbH, Günzburg
  - Nycomed Deutschland GmbH, Gütersloh
  - Nycomed Deutschland GmbH, Haar
  - Nycomed Deutschland GmbH, Hadmersleben
  - Nycomed Deutschland GmbH, Hagen
  - Nycomed Deutschland GmbH, Haigerloch
  - Nycomed Deutschland GmbH, Halbe
  - Nycomed Deutschland GmbH, Halberstadt
  - Nycomed Deutschland GmbH, Haldensleben I
  - Nycomed Deutschland GmbH, Halle
  - Nycomed Deutschland GmbH, Hamburg
  - Nycomed Deutschland GmbH, Hamelin
  - Nycomed Deutschland GmbH, Hanover
  - Nycomed Deutschland GmbH, Haren
  - Nycomed Deutschland GmbH, Harsefeld
  - Nycomed Deutschland GmbH, Hasbergen
  - Nycomed Deutschland GmbH, Haselünne
  - Nycomed Deutschland GmbH, Haunsheim
  - Nycomed Deutschland GmbH, Haßfurt
  - Nycomed Deutschland GmbH, Haßloch
  - Nycomed Deutschland GmbH, Haßmersheim
  - Nycomed Deutschland GmbH, Heddesheim
  - Nycomed Deutschland GmbH, Heek
  - Nycomed Deutschland GmbH, Heide
  - Nycomed Deutschland GmbH, Heidelberg
  - Nycomed Deutschland GmbH, Heidelberg (Boxberg)
  - Nycomed Deutschland GmbH, Heidenheim
  - Nycomed Deutschland GmbH, Heilbronn
  - Nycomed Deutschland GmbH, Heiligenhafen
  - Nycomed Deutschland GmbH, Helmstedt
  - Nycomed Deutschland GmbH, Hemmoor
  - Nycomed Deutschland GmbH, Hennickendorf
  - Nycomed Deutschland GmbH, Hennigsdorf
  - Nycomed Deutschland GmbH, Herbertingen
  - Nycomed Deutschland GmbH, Herbsleben
  - Nycomed Deutschland GmbH, Herdorf
  - Nycomed Deutschland GmbH, Herford
  - Nycomed Deutschland GmbH, Hermsdorf
  - Nycomed Deutschland GmbH, Herne
  - Nycomed Deutschland GmbH, Heroldsberg
  - Nycomed Deutschland GmbH, Herrenberg
  - Nycomed Deutschland GmbH, Herten
  - Nycomed Deutschland GmbH, Herzogenaurach
  - Nycomed Deutschland GmbH, Hessisch Lichtenau
  - Nycomed Deutschland GmbH, Heubach
  - Nycomed Deutschland GmbH, Hildburghausen
  - Nycomed Deutschland GmbH, Hildesheim
  - Nycomed Deutschland GmbH, Hille
  - Nycomed Deutschland GmbH, Hilpoltstein
  - Nycomed Deutschland GmbH, Hirschaid
  - Nycomed Deutschland GmbH, Hirschberg
  - Nycomed Deutschland GmbH, Hofbieber
  - Nycomed Deutschland GmbH, Hohenroth
  - Nycomed Deutschland GmbH, Hollenstedt
  - Nycomed Deutschland GmbH, Holzgerlingen
  - Nycomed Deutschland GmbH, Horb
  - Nycomed Deutschland GmbH, Höchheim
  - Nycomed Deutschland GmbH, Hückelhoven
  - Nycomed Deutschland GmbH, Hüllhorst
  - Nycomed Deutschland GmbH, Ibbenbueren
  - Nycomed Deutschland GmbH, Ifta
  - Nycomed Deutschland GmbH, Igersheim
  - Nycomed Deutschland GmbH, Ilmenau
  - Nycomed Deutschland GmbH, Ilsenburg
  - Nycomed Deutschland GmbH, Ilsfeld
  - Nycomed Deutschland GmbH, Ilvesheim
  - Nycomed Deutschland GmbH, Ingelheim
  - Nycomed Deutschland GmbH, Ingolstadt
  - Nycomed Deutschland GmbH, Iserlohn
  - Nycomed Deutschland GmbH, Isernhagen-Süd
  - Nycomed Deutschland GmbH, Ispringen
  - Nycomed Deutschland GmbH, Itzehoe
  - Nycomed Deutschland GmbH, Jarmen
  - Nycomed Deutschland GmbH, Jembke
  - Nycomed Deutschland GmbH, Jena
  - Nycomed Deutschland GmbH, Jerichow
  - Nycomed Deutschland GmbH, Jesewitz
  - Nycomed Deutschland GmbH, Jettingen
  - Nycomed Deutschland GmbH, Jetzendorf
  - Nycomed Deutschland GmbH, Jockgrim
  - Nycomed Deutschland GmbH, Johanngeorgenstadt
  - Nycomed Deutschland GmbH, Jördenstorf
  - Nycomed Deutschland GmbH, Jübek
  - Nycomed Deutschland GmbH, Jüterbog
  - Nycomed Deutschland GmbH, Kamenz
  - Nycomed Deutschland GmbH, Kamp-Lintfort
  - Nycomed Deutschland GmbH, Kandern
  - Nycomed Deutschland GmbH, Kappeln
  - Nycomed Deutschland GmbH, Karlshuld
  - Nycomed Deutschland GmbH, Karlsruhe
  - Nycomed Deutschland GmbH, Karstädt
  - Nycomed Deutschland GmbH, Katzenelnbogen
  - Nycomed Deutschland GmbH, Katzhütte
  - Nycomed Deutschland GmbH, Kelkheim
  - Nycomed Deutschland GmbH, Keltern
  - Nycomed Deutschland GmbH, Kemnitz
  - Nycomed Deutschland GmbH, Kempenich
  - Nycomed Deutschland GmbH, Kerpen
  - Nycomed Deutschland GmbH, Kiel
  - Nycomed Deutschland GmbH, Kindsbach
  - Nycomed Deutschland GmbH, Kirchberg
  - Nycomed Deutschland GmbH, Kirchehrenbach
  - Nycomed Deutschland GmbH, Kirchheimbolanden
  - Nycomed Deutschland GmbH, Kleve
  - Nycomed Deutschland GmbH, Klingenberg
  - Nycomed Deutschland GmbH, Klingenthal
  - Nycomed Deutschland GmbH, Koblenz
  - Nycomed Deutschland GmbH, Kolitzheim
  - Nycomed Deutschland GmbH, Konstanz
  - Nycomed Deutschland GmbH, Kornwestheim
  - Nycomed Deutschland GmbH, Koßdorf
  - Nycomed Deutschland GmbH, Königs Wusterhausen
  - Nycomed Deutschland GmbH, Königswartha
  - Nycomed Deutschland GmbH, Kösching
  - Nycomed Deutschland GmbH, Köthen
  - Nycomed Deutschland GmbH, Krauschwitz
  - Nycomed Deutschland GmbH, Krefeld
  - Nycomed Deutschland GmbH, Kremmen
  - Nycomed Deutschland GmbH, Kronach
  - Nycomed Deutschland GmbH, Krumpa
  - Nycomed Deutschland GmbH, Kusel
  - Nycomed Deutschland GmbH, Kusterdingen
  - Nycomed Deutschland GmbH, Kühbach
  - Nycomed Deutschland GmbH, Künzelsau
  - Nycomed Deutschland GmbH, Kürten
  - Nycomed Deutschland GmbH, Laatzen
  - Nycomed Deutschland GmbH, Laboe
  - Nycomed Deutschland GmbH, Lampertheim
  - Nycomed Deutschland GmbH, Landau
  - Nycomed Deutschland GmbH, Landshut
  - Nycomed Deutschland GmbH, Langelsheim
  - Nycomed Deutschland GmbH, Langenberg
  - Nycomed Deutschland GmbH, Langenfeld
  - Nycomed Deutschland GmbH, Langenhagen
  - Nycomed Deutschland GmbH, Lappersdorf
  - Nycomed Deutschland GmbH, Lauenburg
  - Nycomed Deutschland GmbH, Lauf
  - Nycomed Deutschland GmbH, Laufenburg
  - Nycomed Deutschland GmbH, Lauingen
  - Nycomed Deutschland GmbH, Lauterbach
  - Nycomed Deutschland GmbH, Lebach
  - Nycomed Deutschland GmbH, Lebus
  - Nycomed Deutschland GmbH, Lehesten
  - Nycomed Deutschland GmbH, Leimen
  - Nycomed Deutschland GmbH, Leinefelde
  - Nycomed Deutschland GmbH, Leingarten
  - Nycomed Deutschland GmbH, Leipheim
  - Nycomed Deutschland GmbH, Leipzig
  - Nycomed Deutschland GmbH, Leisnig
  - Nycomed Deutschland GmbH, Lengerich
  - Nycomed Deutschland GmbH, Lensahn
  - Nycomed Deutschland GmbH, Leubnitz
  - Nycomed Deutschland GmbH, Leutenberg
  - Nycomed Deutschland GmbH, Leutkirch
  - Nycomed Deutschland GmbH, Leverkusen
  - Nycomed Deutschland GmbH, Lichtenfels
  - Nycomed Deutschland GmbH, Limburgerhof
  - Nycomed Deutschland GmbH, Lingen
  - Nycomed Deutschland GmbH, Linnich
  - Nycomed Deutschland GmbH, Lohmen
  - Nycomed Deutschland GmbH, Lommatzsch
  - Nycomed Deutschland GmbH, Lotte
  - Nycomed Deutschland GmbH, Loxstedt
  - Nycomed Deutschland GmbH, Löbejün
  - Nycomed Deutschland GmbH, Löcknitz
  - Nycomed Deutschland GmbH, Löhne
  - Nycomed Deutschland GmbH, Löwenberger Land
  - Nycomed Deutschland GmbH, Lubin
  - Nycomed Deutschland GmbH, Luckenwalde
  - Nycomed Deutschland GmbH, Ludwigsburg
  - Nycomed Deutschland GmbH, Ludwigshafen
  - Nycomed Deutschland GmbH, Lübeck
  - Nycomed Deutschland GmbH, Lüdenscheid
  - Nycomed Deutschland GmbH, Lühmannsdorf
  - Nycomed Deutschland GmbH, Lünen
  - Nycomed Deutschland GmbH, Lütjenburg
  - Nycomed Deutschland GmbH, Lützen
  - Nycomed Deutschland GmbH, Magdeburg
  - Nycomed Deutschland GmbH, Maintal
  - Nycomed Deutschland GmbH, Mainz
  - Nycomed Deutschland GmbH, Mannheim
  - Nycomed Deutschland GmbH, Mansfeld
  - Nycomed Deutschland GmbH, Marburg
  - Nycomed Deutschland GmbH, Marienberg
  - Nycomed Deutschland GmbH, Markkleeberg
  - Nycomed Deutschland GmbH, Markranstädt
  - Nycomed Deutschland GmbH, Marl
  - Nycomed Deutschland GmbH, Marne
  - Nycomed Deutschland GmbH, Massenhausen
  - Nycomed Deutschland GmbH, Märkisch Buchholz
  - Nycomed Deutschland GmbH, Meckenheim
  - Nycomed Deutschland GmbH, Meeder
  - Nycomed Deutschland GmbH, Mendig
  - Nycomed Deutschland GmbH, Menteroda
  - Nycomed Deutschland GmbH, Mering
  - Nycomed Deutschland GmbH, Merseburg
  - Nycomed Deutschland GmbH, Merzen
  - Nycomed Deutschland GmbH, Merzhausen
  - Nycomed Deutschland GmbH, Merzig
  - Nycomed Deutschland GmbH, Messkirch
  - Nycomed Deutschland GmbH, Mettlach
  - Nycomed Deutschland GmbH, Metzingen
  - Nycomed Deutschland GmbH, Meßstetten
  - Nycomed Deutschland GmbH, Miesbach
  - Nycomed Deutschland GmbH, Mildstedt
  - Nycomed Deutschland GmbH, Minden
  - Nycomed Deutschland GmbH, Mittelschmalkalden
  - Nycomed Deutschland GmbH, Moers
  - Nycomed Deutschland GmbH, Monheim
  - Nycomed Deutschland GmbH, Moormerland
  - Nycomed Deutschland GmbH, Moosburg
  - Nycomed Deutschland GmbH, Mosbach
  - Nycomed Deutschland GmbH, Mosbach-Lohrbach
  - Nycomed Deutschland GmbH, Möhlau
  - Nycomed Deutschland GmbH, Mölln
  - Nycomed Deutschland GmbH, Mönchengladbach
  - Nycomed Deutschland GmbH, Mudau
  - Nycomed Deutschland GmbH, Mudersbach
  - Nycomed Deutschland GmbH, Murnau am Staffelsee
  - Nycomed Deutschland GmbH, Murrhardt
  - Nycomed Deutschland GmbH, Mücheln
  - Nycomed Deutschland GmbH, Mühlacker
  - Nycomed Deutschland GmbH, Mühlberg
  - Nycomed Deutschland GmbH, Mühlhausen
  - Nycomed Deutschland GmbH, Mühltroff
  - Nycomed Deutschland GmbH, Mülheim
  - Nycomed Deutschland GmbH, Müncheberg
  - Nycomed Deutschland GmbH, München
  - Nycomed Deutschland GmbH, Münchweiler
  - Nycomed Deutschland GmbH, Münster
  - Nycomed Deutschland GmbH, Münzenberg
  - Nycomed Deutschland GmbH, Nassau
  - Nycomed Deutschland GmbH, Nastätten
  - Nycomed Deutschland GmbH, Nauen
  - Nycomed Deutschland GmbH, Naumburg
  - Nycomed Deutschland GmbH, Neckargemünd
  - Nycomed Deutschland GmbH, Nellingen
  - Nycomed Deutschland GmbH, Nettersheim
  - Nycomed Deutschland GmbH, Nettetal
  - Nycomed Deutschland GmbH, Neu Wulmstorf
  - Nycomed Deutschland GmbH, Neu-Ulm
  - Nycomed Deutschland GmbH, Neubrandenburg
  - Nycomed Deutschland GmbH, Neubrunn
  - Nycomed Deutschland GmbH, Neuendettelsau
  - Nycomed Deutschland GmbH, Neuenkirchen-Vörden
  - Nycomed Deutschland GmbH, Neuhof
  - Nycomed Deutschland GmbH, Neukirch
  - Nycomed Deutschland GmbH, Neuler
  - Nycomed Deutschland GmbH, Neumünster
  - Nycomed Deutschland GmbH, Neunkirchen
  - Nycomed Deutschland GmbH, Neuruppin
  - Nycomed Deutschland GmbH, Neusalza-Spremberg
  - Nycomed Deutschland GmbH, Neusäß
  - Nycomed Deutschland GmbH, Neuss
  - Nycomed Deutschland GmbH, Neustadt
  - Nycomed Deutschland GmbH, Neuwied
  - Nycomed Deutschland GmbH, Niederlehme
  - Nycomed Deutschland GmbH, Nienburg
  - Nycomed Deutschland GmbH, Norderstedt
  - Nycomed Deutschland GmbH, Nordheim
  - Nycomed Deutschland GmbH, Nuremberg
  - Nycomed Deutschland GmbH, Nünchritz
  - Nycomed Deutschland GmbH, Oberaurach
  - Nycomed Deutschland GmbH, Obergünzburg
  - Nycomed Deutschland GmbH, Oberhausen
  - Nycomed Deutschland GmbH, Oberkirch
  - Nycomed Deutschland GmbH, Oberstdorf
  - Nycomed Deutschland GmbH, Obertshausen
  - Nycomed Deutschland GmbH, Oberursel
  - Nycomed Deutschland GmbH, Ochtendung
  - Nycomed Deutschland GmbH, Oderwitz
  - Nycomed Deutschland GmbH, Oelsnitz
  - Nycomed Deutschland GmbH, Oer-Erkenschwick
  - Nycomed Deutschland GmbH, Offenburg
  - Nycomed Deutschland GmbH, Oftersheim
  - Nycomed Deutschland GmbH, Olbernhau
  - Nycomed Deutschland GmbH, Olbersdorf
  - Nycomed Deutschland GmbH, Osloß
  - Nycomed Deutschland GmbH, Osnabrück
  - Nycomed Deutschland GmbH, Ostbevern
  - Nycomed Deutschland GmbH, Osterburg
  - Nycomed Deutschland GmbH, Osterode
  - Nycomed Deutschland GmbH, Ostrach
  - Nycomed Deutschland GmbH, Ostrhauderfehn
  - Nycomed Deutschland GmbH, Otterndorf
  - Nycomed Deutschland GmbH, Ottweiler
  - Nycomed Deutschland GmbH, Östringen
  - Nycomed Deutschland GmbH, Paderborn
  - Nycomed Deutschland GmbH, Panketal
  - Nycomed Deutschland GmbH, Papenburg
  - Nycomed Deutschland GmbH, Parsberg
  - Nycomed Deutschland GmbH, Pasewalk
  - Nycomed Deutschland GmbH, Passau
  - Nycomed Deutschland GmbH, Peine
  - Nycomed Deutschland GmbH, Penig
  - Nycomed Deutschland GmbH, Perl
  - Nycomed Deutschland GmbH, Pfaffenhofen
  - Nycomed Deutschland GmbH, Pforzheim
  - Nycomed Deutschland GmbH, Pfullendorf
  - Nycomed Deutschland GmbH, Pfullingen
  - Nycomed Deutschland GmbH, Pfungstadt
  - Nycomed Deutschland GmbH, Pirmasens
  - Nycomed Deutschland GmbH, Pirna
  - Nycomed Deutschland GmbH, Plauen
  - Nycomed Deutschland GmbH, Pockau
  - Nycomed Deutschland GmbH, Pohlheim
  - Nycomed Deutschland GmbH, Polch
  - Nycomed Deutschland GmbH, Potsdam
  - Nycomed Deutschland GmbH, Preetz
  - Nycomed Deutschland GmbH, Prüm
  - Nycomed Deutschland GmbH, Pullach
  - Nycomed Deutschland GmbH, Pulsnitz
  - Nycomed Deutschland GmbH, Radeberg
  - Nycomed Deutschland GmbH, Radebeul
  - Nycomed Deutschland GmbH, Raisdorf
  - Nycomed Deutschland GmbH, Rastatt
  - Nycomed Deutschland GmbH, Ratingen
  - Nycomed Deutschland GmbH, Reckendorf
  - Nycomed Deutschland GmbH, Regensburg
  - Nycomed Deutschland GmbH, Reichenbach
  - Nycomed Deutschland GmbH, Reilingen
  - Nycomed Deutschland GmbH, Reinsdorf
  - Nycomed Deutschland GmbH, Rellingen
  - Nycomed Deutschland GmbH, Remscheid
  - Nycomed Deutschland GmbH, Rendsburg
  - Nycomed Deutschland GmbH, Reutlingen
  - Nycomed Deutschland GmbH, Rinchnach
  - Nycomed Deutschland GmbH, Rinteln
  - Nycomed Deutschland GmbH, Rippien
  - Nycomed Deutschland GmbH, Rohrbach
  - Nycomed Deutschland GmbH, Rosenfeld
  - Nycomed Deutschland GmbH, Rosengarten
  - Nycomed Deutschland GmbH, Rostock
  - Nycomed Deutschland GmbH, Rotenburg (Wümme)
  - Nycomed Deutschland GmbH, Rottach-Egern
  - Nycomed Deutschland GmbH, Rottenburg
  - Nycomed Deutschland GmbH, Roßbach
  - Nycomed Deutschland GmbH, Rödermark
  - Nycomed Deutschland GmbH, Röhrmoos
  - Nycomed Deutschland GmbH, Röthenbach
  - Nycomed Deutschland GmbH, Rudolstadt
  - Nycomed Deutschland GmbH, Ruhmannsfelden
  - Nycomed Deutschland GmbH, Rutesheim
  - Nycomed Deutschland GmbH, Rühen
  - Nycomed Deutschland GmbH, Rülzheim
  - Nycomed Deutschland GmbH, Saalfeld
  - Nycomed Deutschland GmbH, Saarbrücken
  - Nycomed Deutschland GmbH, Saarlouis
  - Nycomed Deutschland GmbH, Saint Blasien
  - Nycomed Deutschland GmbH, Saint Georgen
  - Nycomed Deutschland GmbH, Saint Wendel
  - Nycomed Deutschland GmbH, Salzgitter
  - Nycomed Deutschland GmbH, Salzhemmendorf
  - Nycomed Deutschland GmbH, Salzmünde
  - Nycomed Deutschland GmbH, Salzwedel
  - Nycomed Deutschland GmbH, Sand
  - Nycomed Deutschland GmbH, Sandesneben
  - Nycomed Deutschland GmbH, Sangerhausen
  - Nycomed Deutschland GmbH, Sarstedt
  - Nycomed Deutschland GmbH, Sayda
  - Nycomed Deutschland GmbH, Scharbeutz
  - Nycomed Deutschland GmbH, Schellerten
  - Nycomed Deutschland GmbH, Schifferstadt
  - Nycomed Deutschland GmbH, Schiffweiler
  - Nycomed Deutschland GmbH, Schkeuditz
  - Nycomed Deutschland GmbH, Schleswig
  - Nycomed Deutschland GmbH, Schliersee
  - Nycomed Deutschland GmbH, Schmalkalden
  - Nycomed Deutschland GmbH, Schmiedeberg
  - Nycomed Deutschland GmbH, Schonungen
  - Nycomed Deutschland GmbH, Schortens
  - Nycomed Deutschland GmbH, Schönberg
  - Nycomed Deutschland GmbH, Schönwalde-Glien
  - Nycomed Deutschland GmbH, Schriesheim
  - Nycomed Deutschland GmbH, Schwabach
  - Nycomed Deutschland GmbH, Schwalmstadt
  - Nycomed Deutschland GmbH, Schwangau
  - Nycomed Deutschland GmbH, Schwanstetten
  - Nycomed Deutschland GmbH, Schwarmstedt
  - Nycomed Deutschland GmbH, Schwarzenberg
  - Nycomed Deutschland GmbH, Schwarzheide
  - Nycomed Deutschland GmbH, Schwäbisch Hall
  - Nycomed Deutschland GmbH, Schwedt
  - Nycomed Deutschland GmbH, Schweinfurt
  - Nycomed Deutschland GmbH, Schwelm
  - Nycomed Deutschland GmbH, Schwerin
  - Nycomed Deutschland GmbH, Schwerte
  - Nycomed Deutschland GmbH, Schwetzingen
  - Nycomed Deutschland GmbH, Seehausen
  - Nycomed Deutschland GmbH, Selm
  - Nycomed Deutschland GmbH, Siegen
  - Nycomed Deutschland GmbH, Sigmaringendorf
  - Nycomed Deutschland GmbH, Silberhausen
  - Nycomed Deutschland GmbH, Silbitz
  - Nycomed Deutschland GmbH, Simonswald
  - Nycomed Deutschland GmbH, Sindelfingen
  - Nycomed Deutschland GmbH, Sinsheim
  - Nycomed Deutschland GmbH, Sittensen
  - Nycomed Deutschland GmbH, Sommerhausen
  - Nycomed Deutschland GmbH, Sondershausen
  - Nycomed Deutschland GmbH, Sömmerda
  - Nycomed Deutschland GmbH, Spaichingen
  - Nycomed Deutschland GmbH, Speyer
  - Nycomed Deutschland GmbH, Spiesen-Elversberg
  - Nycomed Deutschland GmbH, Spremberg
  - Nycomed Deutschland GmbH, Springe
  - Nycomed Deutschland GmbH, Sprockhövel
  - Nycomed Deutschland GmbH, St. Peter
  - Nycomed Deutschland GmbH, Stadthagen
  - Nycomed Deutschland GmbH, Starnberg
  - Nycomed Deutschland GmbH, Stavenhagen
  - Nycomed Deutschland GmbH, Steigra
  - Nycomed Deutschland GmbH, Steinfeld
  - Nycomed Deutschland GmbH, Steinfurt
  - Nycomed Deutschland GmbH, Steinhagen
  - Nycomed Deutschland GmbH, Stendal
  - Nycomed Deutschland GmbH, Stockach
  - Nycomed Deutschland GmbH, Stockelsdorf
  - Nycomed Deutschland GmbH, Stralsund
  - Nycomed Deutschland GmbH, Strausberg
  - Nycomed Deutschland GmbH, Stuhr
  - Nycomed Deutschland GmbH, Stuttgart
  - Nycomed Deutschland GmbH, Suhl
  - Nycomed Deutschland GmbH, Sulingen
  - Nycomed Deutschland GmbH, Sulzbach
  - Nycomed Deutschland GmbH, Sulzfeld
  - Nycomed Deutschland GmbH, Sulzheim
  - Nycomed Deutschland GmbH, Sundern
  - Nycomed Deutschland GmbH, Sülz
  - Nycomed Deutschland GmbH, Tangerhütte
  - Nycomed Deutschland GmbH, Tarp
  - Nycomed Deutschland GmbH, Taucha
  - Nycomed Deutschland GmbH, Teltow
  - Nycomed Deutschland GmbH, Templin
  - Nycomed Deutschland GmbH, Tessin
  - Nycomed Deutschland GmbH, Teterow
  - Nycomed Deutschland GmbH, Themar
  - Nycomed Deutschland GmbH, Tholey
  - Nycomed Deutschland GmbH, Thurnau
  - Nycomed Deutschland GmbH, Torgelow
  - Nycomed Deutschland GmbH, Traunreut
  - Nycomed Deutschland GmbH, Triebes
  - Nycomed Deutschland GmbH, Triptis
  - Nycomed Deutschland GmbH, Troisdorf
  - Nycomed Deutschland GmbH, Trossingen
  - Nycomed Deutschland GmbH, Tutow
  - Nycomed Deutschland GmbH, Tübingen
  - Nycomed Deutschland GmbH, Ueckermünde
  - Nycomed Deutschland GmbH, Uedem
  - Nycomed Deutschland GmbH, Uelsen
  - Nycomed Deutschland GmbH, Uelzen
  - Nycomed Deutschland GmbH, Uffing
  - Nycomed Deutschland GmbH, Ulm
  - Nycomed Deutschland GmbH, Umkirch
  - Nycomed Deutschland GmbH, Unterhaching
  - Nycomed Deutschland GmbH, Unterkirnach
  - Nycomed Deutschland GmbH, Unterwellenborn
  - Nycomed Deutschland GmbH, Überlingen
  - Nycomed Deutschland GmbH, Vaihingen
  - Nycomed Deutschland GmbH, Vallendar
  - Nycomed Deutschland GmbH, Varel
  - Nycomed Deutschland GmbH, Veilsdorf
  - Nycomed Deutschland GmbH, Verden an der Aller
  - Nycomed Deutschland GmbH, Veringenstadt
  - Nycomed Deutschland GmbH, Vierkirchen
  - Nycomed Deutschland GmbH, Viersen
  - Nycomed Deutschland GmbH, Villingen-Schwenningen
  - Nycomed Deutschland GmbH, Visbek
  - Nycomed Deutschland GmbH, Visselhövede
  - Nycomed Deutschland GmbH, Vitzenburg
  - Nycomed Deutschland GmbH, Vöhrenbach
  - Nycomed Deutschland GmbH, Waghäusel
  - Nycomed Deutschland GmbH, Waiblingen
  - Nycomed Deutschland GmbH, Waidhaus
  - Nycomed Deutschland GmbH, Wain
  - Nycomed Deutschland GmbH, Waldbröl
  - Nycomed Deutschland GmbH, Waldbrunn-Strümpfelbrunn
  - Nycomed Deutschland GmbH, Waldshut-Tiengen
  - Nycomed Deutschland GmbH, Walldorf
  - Nycomed Deutschland GmbH, Wallertheim
  - Nycomed Deutschland GmbH, Walschleben
  - Nycomed Deutschland GmbH, Wanzleben
  - Nycomed Deutschland GmbH, Warstein
  - Nycomed Deutschland GmbH, Wattenheim
  - Nycomed Deutschland GmbH, Wedel
  - Nycomed Deutschland GmbH, Weeze
  - Nycomed Deutschland GmbH, Wegeleben
  - Nycomed Deutschland GmbH, Weida
  - Nycomed Deutschland GmbH, Weiden
  - Nycomed Deutschland GmbH, Weil am Rhein
  - Nycomed Deutschland GmbH, Weilheim
  - Nycomed Deutschland GmbH, Weingarten
  - Nycomed Deutschland GmbH, Weinheim
  - Nycomed Deutschland GmbH, Weinsberg
  - Nycomed Deutschland GmbH, Weißenburg
  - Nycomed Deutschland GmbH, Weißenfels
  - Nycomed Deutschland GmbH, Weißenhorn
  - Nycomed Deutschland GmbH, Weißwasser
  - Nycomed Deutschland GmbH, Welbsleben
  - Nycomed Deutschland GmbH, Welden
  - Nycomed Deutschland GmbH, Welver
  - Nycomed Deutschland GmbH, Wennigsen
  - Nycomed Deutschland GmbH, Wenningstedt-Braderup
  - Nycomed Deutschland GmbH, Werne
  - Nycomed Deutschland GmbH, Wernigerode
  - Nycomed Deutschland GmbH, Wesseling
  - Nycomed Deutschland GmbH, Westerrönfeld
  - Nycomed Deutschland GmbH, Wetter
  - Nycomed Deutschland GmbH, Wettringen
  - Nycomed Deutschland GmbH, Weyhe OT Leeste
  - Nycomed Deutschland GmbH, Wickede
  - Nycomed Deutschland GmbH, Wiesbaden
  - Nycomed Deutschland GmbH, Wiesloch
  - Nycomed Deutschland GmbH, Wiggensbach
  - Nycomed Deutschland GmbH, Wilhelmsdorf
  - Nycomed Deutschland GmbH, Wilhelmshaven
  - Nycomed Deutschland GmbH, Wilhermsdorf
  - Nycomed Deutschland GmbH, Willich
  - Nycomed Deutschland GmbH, Wismar
  - Nycomed Deutschland GmbH, Wismar-Wendorf
  - Nycomed Deutschland GmbH, Witten
  - Nycomed Deutschland GmbH, Wittenberg
  - Nycomed Deutschland GmbH, Wittgensdorf
  - Nycomed Deutschland GmbH, Wittstock
  - Nycomed Deutschland GmbH, Witzenhausen
  - Nycomed Deutschland GmbH, Wolfsburg
  - Nycomed Deutschland GmbH, Woltersdorf
  - Nycomed Deutschland GmbH, Worbis
  - Nycomed Deutschland GmbH, Worms
  - Nycomed Deutschland GmbH, Wöbbelin
  - Nycomed Deutschland GmbH, Wörrstadt
  - Nycomed Deutschland GmbH, Wörth
  - Nycomed Deutschland GmbH, Wriedel
  - Nycomed Deutschland GmbH, Wuelfrath
  - Nycomed Deutschland GmbH, Wuppertal
  - Nycomed Deutschland GmbH, Zarrentin
  - Nycomed Deutschland GmbH, Zeil
  - Nycomed Deutschland GmbH, Zeitz
  - Nycomed Deutschland GmbH, Zorge
  - Nycomed Deutschland GmbH, Zschepplin
  - Nycomed Deutschland GmbH, Zschopau
  - Nycomed Deutschland GmbH, Zweibrücken
  - Nycomed Deutschland GmbH, Zwickau
  - Nycomed Deutschland GmbH, Zwiesel

RESULTS

PARTICIPANT FLOW:
Groups:
- Pantoprazole: All patients enrolled
Period: Overall Study
Arm/Group | Pantoprazole
Started | 8616
Completed | 8554
Not Completed | 62
Not completed — Lost to Follow-up | 62

BASELINE CHARACTERISTICS:
Arm/Group | Pantoprazole
Number analyzed (Participants) | 8616
Age Continuous [Mean (Standard Deviation); unit: years] — The measured value is related to the number of 8502 subjects (= valid cases). This number differs from the overall number of baseline participants due to missing data for 114 subjects.
  years | 55.7 (14.51)
Sex/Gender, Customized [Number; unit: percentage of participants]
  Female | 47.8
  Male | 51.7
  Missing data | 0.5
Nicotine use [Number; unit: percentage of participants]
  Smoker | 35.2
  Non-smoker | 64.1
  Missing data | 0.7
Alcohol use [Number; unit: percentage of participants]
  Daily | 22.1
  Not daily | 77.2
  Missing data | 0.8
Drug abuse [Number; unit: percentage of participants]
  Drug abuse | 2.9
  No drug abuse | 96.0
  Missing data | 1.1
Indication for prescription of pantoprazole [Number; unit: percentage of participants]
  long-term therapy and/or relapse prophylaxis | 50.5
  Acute reflux oesophagitis | 49.1
  Missing data | 0.4

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Severity of Sleep Disturbances
Description: Physician's assessment on a scale with 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: first and last visit (after a median of 18 days)
Population: All patients included and treated, intention to treat, missing values not imputed
Measure: Number; unit: percentage of participants
Groups:
- Pantoprazole / Start of Therapy; Pantoprazole / End of Therapy: All patients with valid values ('as observed')
Arm/Group | Pantoprazole / Start of Therapy | Pantoprazole / End of Therapy
Number analyzed (Participants) | 8616 | 8616
percentage of participants
  None | 13.8 | 77.4
  Mild | 38.2 | 20.0
  Moderate | 35.9 | 1.1
  Severe | 8.0 | 0.07
  Missing data | 4.1 | 1.4

2. Primary Outcome: Assessment of Change of Quality of Sleep During Therapy With Pantoprazole
Description: Physician's assessment on a scale with
  * considerably improved
  * improved
  * unchanged
Time Frame: last visit (after a median of 18 days)
Population: All patients included and treated, intention to treat, missing values not imputed
Measure: Number; unit: percentage of participants
Groups:
- Pantoprazole: All patients with valid values ('as observed')
Arm/Group | Pantoprazole
Number analyzed (Participants) | 8616
percentage of participants
  Considerably improved | 56.2
  Improved | 25.7
  Unchanged | 13.5
  Missing data | 4.6

3. Secondary Outcome: Assessment of the Severity of Heartburn
Description: Physician's assessment on a scale with 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: first and last visit (after a median of 18 days)
Population: Patients included and treated with valid data at first and last visit (without imputation of missing values), intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pantoprazole: All patients with valid values at first and last visit
Arm/Group | Pantoprazole
Number analyzed (Participants) | 8540
units on a scale
  Start of therapy | 3.04 (0.79)
  End of study | 1.34 (0.51)

4. Secondary Outcome: Assessment of the Severity of Eructation/Acid Eructation
Description: Physician's assessment on a scale with 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: first and last visit (after a median of 18 days)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 8540
units on a scale
  Start of therapy | 2.66 (0.88)
  End of study | 1.29 (0.49)

5. Secondary Outcome: Assessment of the Severity of Epigastric Complaints/Epigastric Pain
Description: Physician's assessment on a scale with 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: first and last visit (after a median of 18 days)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 8528
units on a scale
  Start of therapy | 2.25 (0.91)
  End of study | 1.18 (0.42)

6. Secondary Outcome: Assessment of the Severity of Sensation of Fullness/Abdominal Distension
Description: Physician's assessment on a scale with 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: first and last visit (after a median of 18 days)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 8516
units on a scale
  Start of therapy | 2.35 (0.95)
  End of study | 1.28 (0.50)

7. Secondary Outcome: Assessment of the Efficacy of Pantoprazole at Final Visit
Description: Physician's assessment on a scale with 1=excellent, 2=good, 3=satisfactory, 4=not satisfactory
Time Frame: last visit (after a median of 18 days)
Population: Patients included and treated with at least one application of pantoprazole (without imputation of missing values), intention to treat
Measure: Number; unit: percentage of participants
Groups:
- Pantoprazole: Patients included and treated with at least one application of pantoprazole
Arm/Group | Pantoprazole
Number analyzed (Participants) | 8616
percentage of participants
  Excellent | 78.1
  Good | 19.6
  Satisfactory | 1.3
  Not satisfactory | 0.2
  Missing data | 0.8

8. Secondary Outcome: Assessment of the Tolerability of Pantoprazole at Final Visit
Description: Physician's assessment on a scale with 1=excellent, 2=good, 3=satisfactory, 4=not satisfactory
Time Frame: last visit (after a median of 18 days)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Pantoprazole
Number analyzed (Participants) | 8616
percentage of participants
  Excellent | 81.6
  Good | 14.8
  Satisfactory | 0.4
  Not satisfactory | 0.06
  Missing data | 3.1

ADVERSE EVENTS:
Time Frame: From first until last visit
Arm/Group | Pantoprazole
Serious Adverse Events (participants affected / at risk) | 2/8616
Other Adverse Events (participants affected / at risk) | 11/8616
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pantoprazole (N=8616)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.01% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pantoprazole (N=8616)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No